CLINICAL TRIAL: NCT07030556
Title: Cascading an Intervention to Promote Healthy Sleep Among Adolescents Following Vocational Education Via a Participatory Approach
Brief Title: Cascading A Healthy Sleep Intervention In Vocational Education
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ONZ-2024-0614
Record Dates: First submitted 2025-06-04; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Sleep Quality; Implementation
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Sleep Intervention (Experimental): This single-arm study involves three interventions: (A) a co-creation process with 6-8 purposefully selected students and teachers to adapt an existing healthy sleep intervention to local needs; (B) a one-time training for teachers on the importance of sleep and implementation of the intervention, supported by thematic manuals and follow-up consultations; and (C) school-wide implementation of the adapted healthy sleep intervention for all first- and second-year secondary students.
  Interventions: Other: Healthy Sleep Intervention; Other: Co-creation process; Other: Training for teachers

INTERVENTIONS:
Other: Healthy Sleep Intervention — This intervention has a duration of nine weeks and starts with a kick-off event where the students of the action group provide explanations to fellow students. Furthermore, the intervention is structured in five themes of approximately two weeks each: 1) importance of healthy sleep, 2) sleep and wake cycle, 3) screen time, 4) exercise and nutrition and 5) screen use and mental well-being. Three posters are provided for each theme, five to seven Instagram posts and a class discussion. In addition, healthy sleep is explained during the biology lesson. Furthermore, a competition between classes is organized to sleep as well as possible with the help of an app, classes are given a planner to visualize the workload of school tasks, exercise snacks will be introduced during the lessons and students are given a notebook to write things down in case of worrying. Finally, a closing moment is provided. Flyers with information about healthy sleep in young people are distributed to parents.
Other: Co-creation process — co-creation process with students and teachers: to adapt the existing intervention to the needs of the school. For this, schools can recruit 6 to 8 students via purposeful sampling to form an action group. They will be asked to participate in two sessions during the lunch break in which 1) the needs of the students at school in relation to healthy sleep are mapped out and the goals of the already developed intervention are supplemented or not based on the needs 2) a choice is made from the already developed intervention components 3) necessary adjustments are made to intervention components.
Other: Training for teachers — implementation of the implementation intervention for teachers. The implementation intervention consists of a one-off training for all teachers of the 1st and 2nd year of secondary school in which the importance of sleep and the intervention and its materials are explained. A manual per theme is then provided to the teachers who will implement components (see also appendix 'Manual Sleep Project'). Consultation moments will be planned in consultation to discuss the progress of the implementation.

SUMMARY:
Sleep is crucial for the mental, cognitive and physical health of adolescents. However, teenagers in 2024 sleep less and less and their sleep is of poorer quality. It is striking that adolescents who follow vocational education sleep even worse compared to peers who follow a technical or general education. It is therefore important to focus on this risk group of adolescents to reduce health differences. However, there are no previous intervention studies that focused on them.

In previous research, a healthy sleep intervention was already developed, implemented and evaluated in a participatory manner. Within this research, the investigators want to focus on evaluating the process of implementation of this intervention among first and second year secondary school students (12 to 14 year olds) and teachers from vocational education. Based on the results of this process evaluation, the investigators want to deliver this intervention as a ready-made package to Flemish secondary schools.

ELIGIBILITY:
Inclusion Criteria:

* student in 1st or 2nd year of secondary vocational education
* teacher who helped implement the intervention

Exclusion Criteria:

* No students who participated in the co-creation process may participate in the group interview about receiving the intervention.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
process evaluation of the implementation of a healthy sleep intervention | From enrollment to the end of intervention implementation at 3 months
  experiences of students with the received intervention; experiences of students and teachers regarding the participatory adaptation of the intervention; experiences of teachers with the implementation of the intervention.
  this will be analysed through interviews and focus groups

CONTACTS AND LOCATIONS:
Overall Officials: Benedicte Deforche, Prof. PhD, Principal Investigator — University Ghent
Locations (1):
- Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No
it is not necessary to share individual participant data as part of a result of this study.